CLINICAL TRIAL: NCT05828420
Title: The Effect of Music the Mother Listened to During Her Pregnancy, White Noise and Heart Sound on Neonatal Pain During Heel Lance
Brief Title: The Effect of Music, White Noise and Heart Sound on Neonatal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Birsen Mutlu, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: bdonmez@iuc.edu.tr
Record Dates: First submitted 2023-02-27; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Neonatal; Pain
Keywords: Music; Neonatal; pain; white noise; heel lance; heart sound
MeSH Terms: conditions — Pain | interventions — Heart Sounds; Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The pain effect of listening to white noise on newborn babies (Experimental): Each baby was listened to white noise 10 minutes before, during and 20 minutes after the painful attempt.
  Interventions: Other: White noise
- The pain effect of listening to heart sound on newborn babies (Experimental): Each baby listened to heart sounds at an average rate of 70 beats 10 minutes before, during and 20 minutes after the painful procedure.
  Interventions: Other: Heart sound
- The pain effect of listening to music on newborn babies (Experimental): Each baby was listened to the music that the mother listened to the most during pregnancy restriction 10 minutes before, during and after the painful attempt.
  Interventions: Other: Music

INTERVENTIONS:
Other: White noise — Each baby was listened to white noise 10 minutes before, during and 20 minutes after the painful attempt.
  Arms: The pain effect of listening to white noise on newborn babies
Other: Heart sound — Each baby listened to heart sounds at an average rate of 70 beats 10 minutes before, during and 20 minutes after the painful procedure.
  Arms: The pain effect of listening to heart sound on newborn babies
Other: Music — Each baby was listened to the music that the mother listened to the most during pregnancy restriction 10 minutes before, during and after the painful attempt.
  Arms: The pain effect of listening to music on newborn babies

SUMMARY:
Infants are exposed to many painful procedures during their stay in the Neonatal Intensive Care Unit (NICU). Some epidemiological studies report that infants experience an average of 7.5-14 painful procedures per day per infant during the first 14 days of their hospitalization.

The most significant problem encountered in understanding pain in infants is the lack of verbal expression of pain. Newborns express their pain with nonverbal behavioral expressions. Therefore, any pain assessment is based on the ability to recognize the pain symptoms of others. The pain experienced may cause physiological imbalances and abnormalities in brain development and stress response in infants in the short and long term. It can negatively affect family-infant communication, as well as cause emotional and psychosomatic problems later in life.

Today, music therapy has positive effects on reducing stress, reducing pain, oxygen saturation level, and peak heart rate values in providing individualized developmental care of the infant in neonatal intensive care units. Heart sound, babies hear the mother's heart sound the most during the intrauterine period in the womb. Therefore, when babies hear the sound, they are familiar with in the womb, they will feel safe and a sense of relaxation will occur in the baby. Several studies have proven that playing heartbeat sounds to newborn babies can positively affect their physiological indicators, feeding, length of hospital stay and pain outcomes. The current literature shows that the presence of rhythmic sound can positively affect the neurobehavioral development of the infant and reduce pain. Rhythmic sounds have healing/positive effects on newborns; listening to white noise reduces preterms' pain scores, stabilizes vital signs, and plays an active role in preterms' sleep-wake period.

In line with all this information, this study was carried out as a randomized controlled experimental study in order to determine the effects of music played during heel spear application, white noise and heart sound in infants.

DETAILED DESCRIPTION:
The purpose of the study is to determine the effect of white noise, heart sound, and music on reducing neonatal pain during heel lance.

The design of the study is a randomized controlled experimental design. The sample of the study consisted of 84 infants with a gestational age of 28-42 weeks. The infants were exposed to white noise, heart sounds, or the music that the mother listened to most frequently during pregnancy for 10 minutes before the heel lance, during, and 20 minutes after the procedure. The pain of the infants before, during, and after the procedure was measured using the Neonatal Infant Acute Pain Assessment Scale (NIAPAS). Also, the duration of the procedure and the crying time were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Having a 28-42 weeks preterm or term newborn
* No sedative or analgesic given in the last 6 hours
* Parental consent for inclusion in the study in line with participant information and consent form.

Exclusion Criteria:

* Presence of intracranial bleeding
* Having cerebral hypoxic ischemia
* Babies whose blood cannot be drawn on the first try

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
NIAPAS pain score | 2 year
  The Neonatal Infant Acute Pain Assessment Scale (NIAPAS) was used to measure the pain of newborns. The score that can be obtained from scoring the indicators is between 0-18. The indicators can be scored with 2 (0,1), 3 (0,1,2) or 4 (0,1,2,3) grades. Painful procedures are evaluated in three stages. Pain intensity is classified as mild (0-5), moderate (6-9), and severe pain (10-18).

SECONDARY OUTCOMES:
Crying time | 2 year
  Infant's crying time were calculated by watching the video recordings. Pain assessment of the infants was performed by two independent neonatal nurses, different from the researcher, by watching the video recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Mutlu, Principal Investigator — İstanbul Universty-Cerrahpaşa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No